CLINICAL TRIAL: NCT06658548
Title: Effects of Isometric Hand Grip Exercise Training on Lung Function in COPD Patients
Brief Title: Isometric Hand Grip Exercise and Lung Function in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hajra Qazi
Record Dates: First submitted 2024-09-16; First posted 2024-10-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary functions; Hand grip strength; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Isometric handgrip exercise training with resistance exercise; Other: Resistance Exercise
- Group B (Active Comparator)
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Isometric handgrip exercise training with resistance exercise — The subjects will perform 24 consecutive days, an isometric handgrip exercise at 30% Maximum Voluntary Contraction (M.V.C)continue the exercise protocol for another 48 consecutive days.
  Arms: Group A
Other: Resistance Exercise — The subjects will undergo outpatient training intervention during a period of 8 weeks will be using a hypertrophic maximum strength training method, which will divided into three phases: (1) muscle habituation training (2 weeks), (2) hypertrophic training I (5 weeks), and (3) hypertrophic training II, with intensified eccentric work (5 weeks).

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a preventable and treatable lung disease. People with COPD must work harder to breathe, which can lead to shortness of breath and/or feeling tired. Early in the disease, people with COPD may feel short of breath when they exercise. As the disease progresses, it can be hard to breathe out (exhale) or even breathe in (inhale). A person with COPD may have obstructive bronchiolitis emphysema, or a combination of both conditions. There is variety of treatment like breathing exercises, inspiratory muscle training exercises, resistance training and aerobic exercise to improve lung function as well as to decrease the chances of cardiopulmonary complications. the purpose of this study it to observe the effects of hand gripping isometric exercises on pulmonary functions in COPD patients.

Study design will be randomized clinical trial in which experiment group will receive isometric training with resistance training and other group will only receive resistance training . Total forty eight participates will recruited with convince sampling, after that we will use simple random sampling to divide the patient into both equal groups. Digital spirometry will be used to document the pulmonary function also to observe the difference in post treatment.Data analysis will be done using SPSS version 25.

DETAILED DESCRIPTION:
The most common respiratory symptoms associated with COPD include dyspnea, cough and/or sputum production. In addition to the daily symptom burden, COPD may be punctuated by periods of acute worsening of respiratory symptoms (often referred to as 'exacerbations'), which account for the greatest proportion of total COPD burden on healthcare systems. COPD can be progressive, as indicated by reductions in spirometry measures such as forced expiratory volume in 1 s (FEV1) over time, though patients may progress at different rates.

Physical exercise is a major component of the total therapeutic regimen in pulmonary rehabilitation and has been positively correlated with better lung function in all age groups. Physical activity may attenuate age-related decline in pulmonary function and should be an integral part of pulmonary rehabilitation to improve lung function. Respiratory diseases constitute a major socioeconomic and a massive health burden all over the world. It represents an enormous drain on human and financial resources, and also contributes largely to morbidity and mortality at both global and national scales.

Age related decline in pulmonary function even in the absence of extrinsic pollutants, which can be caused by several factors related to the lung tissue itself. This age related decline further causes a reduction in exercise capacity and contributes immensely to loss of muscle power and mobility with progressive airflow limitation. The reduction in muscle power and increased airflow limitation contribute to the loss of muscle mass, decreased functional capacity and eventually loss of independence .Handgrip exercises are easy to perform, take less space and are more accessible in various locations such as hospitals, schools, in transit and in the home; therefore, it can lead to increased adherence to treatment.

A good number of scientific studies clearly demonstrate that isometric exercise is efficacious in the attenuation of resting blood pressure in both normotensive and hypertensive subjects. Isometric exercise produced greater reductions in systolic and diastolic blood pressure compared to dynamic exercise training. Moreover, physical exercise has been shown to be a non-pharmacological prophylactic regimen as it is capable of protecting against decline in pulmonary functions due to aging and enhances the physiological responses of the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 40 to 70 years
* Clinical or functional diagnosis of COPD criteria GOLD II and III
* Clinically stable (outside the period of exacerbation of the disease for at least 3 months),
* Independently able to perform instrumental activities of daily living, as assessed by the functional activities questionnaire
* No medical contraindications for physical exercise

Exclusion Criteria:

* Pulmonary diseases such as asthma, pulmonary fibrosis, pneumonia and other non-pulmonary
* Sever or difficult to control ( heart disease or sequelae of acute or chronic orthopedic and/or neurological diseases),
* Those who use walking assist devices that could influence the exercise
* Enrolled in a physical training program within the last 3 months at baseline

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | Baseline; 5th Week; 10th Week
  6MWT is a sub-maximal exercise test used to examine person aerobic capacity and endurance. This test initially developed to make an assessment of patient with cardiopulmonary issues. It is used to check the functional capacity of the individual and it provides useful information regarding all the body systems during physical activity, including cardiovascular and pulmonary system. It can used for all age group range 2 to above 64 years The test is easy to perfume , with standardized limited instructions and encouragement being given as person walk as far as possible over 6 minutes through a flat corridor. The final distance is recorded in meters.
Forced Vital Capacity (FVC) | Baseline; 5th Week; 10th Week
  The FVC is the forced vital capacity. It requires that the subject make a maximal inspiration to TLC, then make a maximal forced expiratory effort, leaving only the RV. In a normal subject, the FEV1/FVC is greater than 0.8; patients with obstructive lung disease, such as asthma or COPD, show a decreased FEV1/FVC
Forced Expiratory Volume in 1 second (FEV1) | Baseline; 5th Week; 10th Week
  Forced expiratory volume (FEV1) calculates the amount of air that a person can force out of their lungs in 1 second. FEV1 values that are lower than average suggest the presence of COPD.
FEV1/FVC Ratio | Baseline; 5th Week; 10th Week
  The FEV1/FVC ratio is a measurement of lung function that compares the forced expiratory volume in one second (FEV1) to the forced vital capacity (FVC). It is used to help diagnose and monitor lung conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fonseca J, Machado FVC, Santin LC, Andrello AC, Schneider LP, Fernandes Belo L, Rodrigues A, Fernandes Rugila D, Furlanetto KC, Hernandes NA, Pitta F. Handgrip Strength as a Reflection of General Muscle Strength in Chronic Obstructive Pulmonary Disease. COPD. 2021 Jun;18(3):299-306. doi: 10.1080/15412555.2021.1919608. Epub 2021 May 7. PMID 33961519
- [Background] Felipe C, Bartolome C, Miguel D, Victor PP. Longitudinal changes in handgrip strength, hyperinflation, and 6-minute walk distance in patients with COPD and a control group. Chest. 2015 Oct;148(4):986-994. doi: 10.1378/chest.14-2878. PMID 25996450
- [Background] Lau CW, Leung SY, Wah SH, Yip CW, Wong WY, Chan KS. Effect on muscle strength after blood flow restriction resistance exercise in early in-patient rehabilitation of post-chronic obstructive pulmonary disease acute exacerbation, a single blinded, randomized controlled study. Chron Respir Dis. 2023 Jan-Dec;20:14799731231211845. doi: 10.1177/14799731231211845. PMID 37976375
- [Background] Kovarik M, Joskova V, Patkova A, Koblizek V, Zadak Z, Hronek M. Hand grip endurance test relates to clinical state and prognosis in COPD patients better than 6-minute walk test distance. Int J Chron Obstruct Pulmon Dis. 2017 Dec 1;12:3429-3435. doi: 10.2147/COPD.S144566. eCollection 2017. PMID 29238187
- [Background] Qiu P, Chen M, Lv S, Xie J, Wu J. The association between walking pace and hand grip strength with the risk of chronic obstructive pulmonary disease: a bidirectional Mendelian randomization study. BMC Pulm Med. 2023 Nov 20;23(1):450. doi: 10.1186/s12890-023-02759-z. PMID 37986176
- [Background] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160